CLINICAL TRIAL: NCT01712971
Title: Reduced Intra-operative Blood Loss in Pancreaticoduodenectomy for Pancreatic or Peri-ampullary Tumors; Monocentric Randomized Trial on Standard Open Versus Minimally Invasive Surgery
Brief Title: Reduced Intra-operative Blood Loss in Pancreaticoduodenectomy for Pancreatic or Peri-ampullary Tumors; Monocentric Trial on Standard Open Versus Minimally Invasive Surgery
Status: Withdrawn | Type: Observational
Sponsor: Baki Topal (Other)
Responsible Party: Sponsor-Investigator, Baki Topal, Professor of Surgery, University Hospital, Gasthuisberg
Organization: University Hospital, Gasthuisberg (Other)
Other Study IDs: LPD
Record Dates: First submitted 2012-10-18; First posted 2012-10-24 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Surgery; Pancreatic Tumour; Peri-ampullary Tumour; Blood Loss
Keywords: surgery; pancreas; tumour; blood loss
MeSH Terms: conditions — Pancreatic Neoplasms; Hemorrhage; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OPD: standard open pancreaticoduodenectomy
- LPD: laparoscopic pancreaticoduodenectomy

SUMMARY:
The incidence of complications after standard open pancreaticoduodenectomy for pancreatic or peri-ampullary tumours is around 50%. The amount of intra-operative blood loss is an important factor that determines the occurrence of postoperative complications. Therefore, any significant reduction of intra-operative blood loss will benefit the peri-operative course.

DETAILED DESCRIPTION:
Pancreaticoduodenectomy (PD) is the only therapeutic option to cure patients suffering from pancreatic head or peri-ampullary tumors. The standard approach in PD is open surgery (OPD). With advancing technology, data from expert centers suggest minimally invasive or laparoscopic PD (LPD) to be safe and feasible, though randomized studies are lacking to show the clinical benefits of LPD vs. OPD.

Advantages of minimally invasive surgery over open surgery are reduced tissue damage, surgical trauma and immunosuppression.

The general objective of this study is to compare the intra-operative efficacy of LPD vs. OPD, and in particular the amount of intra-operative blood loss.

Study design Monocentric randomized trial to compare the amount of intra-operative blood loss in LPD vs. OPD. Patients expected to undergo portal vein resection/reconstruction or any simultaneous other type of surgery will be excluded from the study.

Two experienced surgeons will perform all procedures; RA will perform the open and BT the laparoscopic procedures. A pylorus-resecting PD will be followed by a trans-mesocolic end-to-side hepatico-jejunostomy (HJS), a pancreatico-gastrostomy (PGS), and an ante-colic gastro-enterostomy (GES). Da Vinci robotic assistance of the reconstruction in LPD is allowed for the HJS and the PGS, while the GES will be done with endo-staplers.

Statistical considerations Randomization will take place pre-operatively after informed consent has been obtained. Patients will be randomized into two groups (OPD vs. LPD) using permuted blocks of size 6. This implies that of each series of 6 consecutive patients, three patients will be randomized in each group. There are no stratification variables.

Monocentric randomized trial to compare the amount of intra-operative blood loss in LPD vs. OPD. Patients expected to undergo portal vein resection/reconstruction or any simultaneous other type of surgery will be excluded from the study.

Reference intra-operative blood loss levels are available from 138 patients (June 2009 - June 2012), without portal vein resection and without additional surgery. Analysis of these data reveals that these values follow a lognormal distribution; the log-transformed blood loss has a normal distribution with mean and standard deviation equal to 6.06 and 0.83, respectively. The corresponding geometric mean equals 427ml. Based on this distribution, 42.4%, 24.7% and 15.1% of the subjects are expected to have blood loss higher than 500, 750 and 1000 ml, respectively. It is assumed that the treatment (LPD) will lead to a 50% reduction of the (geometric) mean. The impact of this assumption on the distribution of the blood loss levels implies that 15.1%, 6.4% and 3.1% of the subjects in the LPD-group are expected to have a blood loss level higher than 500, 750 and 1000 ml, respectively.

Based on a two-sided two-sample pooled t-test of a mean ratio with lognormal data, a total of 50 subjects is needed to detect a two-fold reduction in blood loss (with alpha set at 5%) with 90% power.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, who undergo PD for a pancreatic or peri-ampullary tumor
* Age between 18 to 80 years
* Patients with and without pre-operative biliary drainage (for obstructive jaundice)
* Pre-operative radiotherapy, chemotherapy, or biological is allowed
* PD for IPMN is allowed

Exclusion Criteria:

* Planned concomitant surgical procedures such as simultaneous colonic resection etc.
* Expected/planned reconstruction of the portal vein or superior mesenteric vein
* Any arterial reconstruction at the time of surgery
* Age < 18years
* Pregnancy
* PD for chronic pancreatitis
* PD for pancreatic trauma
* PD for post-ERCP complications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from pancreatic or peri-ampullary tumour
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2014-01 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
intra-operative blood loss | day 0 (at the end of surgery)
  the amount of intra-operative blood loss (ml) at the end of surgery (d0)

SECONDARY OUTCOMES:
Surgical resection margin | day 30
  Histopathological examination of surgical resection margins of the resection specimen; done within 30 days after surgery pR0: tumour-free resection margins pR1: tumour involvement of surgical resection margins
length of hospital stay after surgery | day 30; 60; 90; 180
  discharge from hospital after surgery
hospital costs | year 1 & 2
  final cost analysis

CONTACTS AND LOCATIONS:
Overall Officials: Baki Topal, MD, PhD, Study Director — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium